CLINICAL TRIAL: NCT01500343
Title: A Pilot Study of Probiotic Saccharomyces Boulardii Use in Chronic Heart Failure Patients
Brief Title: A Pilot Study of Probiotic Saccharomyces Boulardii Use in Chronic Heart Failure Patients. Estudo PROICA
Acronym: PROICA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Annelise Cisari Costanza, Principal investigator, Universidade Federal Fluminense
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UFF-Cardiologia-01
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Last update posted 2011-12-28 (Estimated); Status verified 2011-12

CONDITIONS: Heart Failure
Keywords: heart failure; probiotics; Saccharomyces boulardii; cardio-intestinal syndrome; gut; inflammation
MeSH Terms: conditions — Heart Failure; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saccharomyces boulardii (Experimental)
  Interventions: Drug: Saccharomyces boulardii
- Placebo (Placebo Comparator)
  Interventions: Drug: Saccharomyces boulardii

INTERVENTIONS:
Drug: Saccharomyces boulardii — 1 gram per day, during 3 months

SUMMARY:
The purpose of this study is to evaluate the feasibility, safety and effects in inflammatory response of the therapy with a probiotic agent, the yeast Saccharomyces boulardii (SB), in chronic heart failure patients.

DETAILED DESCRIPTION:
A cardiointestinal syndrome has been described in heart failure patients, with morphologic and functional intestinal disorders, increased enteropathogenic bacteria concentration, bacterial translocation and inflammatory activation, thus contributing for clinical worsening and progression of the disease.

In clinical practice, probiotics has been used in several different conditions, as inflammatory bowel diseases, acute and antibiotic-associated diarrhea, food allergies, and cancer, showing benefits in inflammation and reducing bacterial translocation. However, the use of probiotics in heart failure has never been described.

ELIGIBILITY:
Inclusion Criteria:

* Class I or II (NYHA)heart failure patients

Exclusion Criteria:

* Corticosteroid use within 30 days
* NSAID use within 30 days
* Antibiotic use within 30 days
* Acute infections
* Inflammatory diseases
* Autoimmune diseases
* Cancer
* Intestinal diseases
* Chronic renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-11; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Analysis of biochemical profile (high-sensitivity C reactive protein, total leukocyte count and uric acid seric levels) | 3 months
  Analysis at baseline and after intervention

SECONDARY OUTCOMES:
Analysis of cardiac remodelling | 3 months
  Ecocardiographic analysis of left atrial diameter and left ventricular ejection fraction at baseline and after intervention
Analysis of creatinine seric levels | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Annelise C Costanza, MD, Principal Investigator — Universidade Federal Fluminense; Evandro T Mesquita, MD,PhD, Study Director — Universidade Federal Fluminense
Locations (1):
- Hospital Universitário Antonio Pedro, Niterói, Rio de Janeiro, Brazil